CLINICAL TRIAL: NCT01021488
Title: Rosuvastatin for Prevention of Deep Vein Thrombosis in Patients Undergoing Total Knee Replacement Arthroplasty: STOP DVT - A Prospective Randomized Controlled Trial
Brief Title: Rosuvastatin for Preventing Deep Vein Thrombosis
Acronym: STOP-DVT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Hallym University Sacred Heart Hospital, Department of Internal Medicine, Division of Cardiology, Hallym University Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009-I053
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2009-11

CONDITIONS: Deep Vein Thrombosis; Venous; Thrombosis; Prevention
Keywords: Thrombosis; Vein; Statin; Prevention
MeSH Terms: conditions — Venous Thrombosis; Thrombosis | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental: Rosuvastatin + enoxaparin arm (Experimental): Rosuvastatin 20mg/day for 7days before and 7days after index surgery (total knee replacement arthroplasty, TKRA) Enoxaparin 40mg SQ/day 12hr before TKRA and from 1day to 7day after TKRA should be administered at the same time with rosuvastatin.
  Interventions: Drug: Rosuvastatin 20mg/d for 14days
- enoxaparin only (Active Comparator): enoxaparin 40mg sq/day only starting 12hr before TKRA and from on day 1 to 7 after index surgery
  Interventions: Drug: enoxaparin only

INTERVENTIONS:
Drug: Rosuvastatin 20mg/d for 14days — Rosuvastatin 20mg/day for 7days before and 7days after index surgery (total knee replacement arthroplasty, TKRA) Enoxaparin 40mg SQ/day 12hr before TKRA and from 1day to 7day after TKRA should be administered at the same time with rosuvastatin.
  Arms: Experimental: Rosuvastatin + enoxaparin arm
Drug: enoxaparin only — enoxaparin 40mg sq/day only starting 12hr before TKRA and from on day 1 to 7 after index surgery
  Arms: enoxaparin only

SUMMARY:
Deep vein thrombosis (DVT)is devastating disease which influencing the mortality and morbidity of patients at-risk like those undergoing orthopedic surgery.

Recent publication suggested HMO-co-A reductase inhibitor (statin) may reduce the occurrence rate of venous thromboembolism in apparently healthy persons.

The pleiotropic property of statin like antioxidant, antithrombotic, anti-inflammatory may have effect on the positive results.

We are investigating whether rosuvastatin is associated with lower incidence of deep vein thrombosis (DVT) in patients undergoing total knee replacement arthroplasty(TKRA)who are at-high risk for developing DVT

ELIGIBILITY:
Inclusion Criteria:

* Patients who are going to receive total knee replacement arthroplasty from any cause.
* < 19 years old

Exclusion Criteria:

* patients with cancer
* Patients receiving anticoagulant agents from any cause
* current statin users
* expecting survival from other co-morbidity < 1year
* Bed ridden patient
* AST, ALT > 3times of upper normal limit
* CK> upper normal limit
* pregnancy
* patients who receives hormone replacement therapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Development of deep vein thrombosis diagnosed and confirmed by CT angiography at lower extremities | 7days after index surgery

SECONDARY OUTCOMES:
D-dimer, lipid panel (Total cholesterol, TG, HDL, LDL), hsCRP, CK, transaminase, ALP | 7days, 1month, 2month after index surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Ho Jo, MD, Principal Investigator — Hallym University Medical Center; Sang-Ho Jo, MD, Study Director — Hallym University Medical Center; Young-Jin Choi, MD, Study Chair — Hallym University Medical Center
Locations (1):
- Hallym University Sacred Heart Hospital, Department of Cardiology and Orthopedic Surgery, Anyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Lippi G, Favaloro EJ, Sanchis-Gomar F. Venous thrombosis associated with HMG-CoA reductase inhibitors. Semin Thromb Hemost. 2013 Jul;39(5):515-32. doi: 10.1055/s-0033-1343892. Epub 2013 Apr 29. PMID 23629822
- [Derived] Park WJ, Jo SH, Kim SA, Kim HS, Han SJ, Choi YJ, Rhim CY. Rationale and design of STOP DVT study: rosuvastatin for the prevention of deep vein thrombosis in patients undergoing total knee replacement arthroplasty--a prospective randomized open-label controlled trial. Contemp Clin Trials. 2011 Sep;32(5):779-82. doi: 10.1016/j.cct.2011.06.001. Epub 2011 Jun 12. PMID 21684353